CLINICAL TRIAL: NCT01942161
Title: A Multicenter, Double-blind, Randomized, Dose-comparison Study of Three Different Doses of Aripiprazole (2 mg/Day, 6-12 mg/Day, 24-30 mg/Day) Orally Administered Over 6 Weeks in Pediatric Patients (Aged 13-17 Years) With Schizophrenia
Brief Title: A Short Treatment Study of Aripiprazole in Pediatric Patients With Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-09-003; JapicCTI-101146 (Other: JAPIC)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia
Keywords: Schyzophrenia, pediatric patients
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low (2 mg/day) (Experimental): Subjects in the 2 mg/day group will be administered 2 mg once daily for 6 weeks (42 days).
  Interventions: Drug: Aripiprazole Low (2 mg/day)
- Mid (6 - 12 mg/day) (Experimental): Subjects in the 6-12 mg/day group will be administered 2 mg once daily for 2 days, followed by a maintenance dose of 6 mg for 40 days. From Day 15 onwards, the dose may be increased to 12 mg in accordance with the criteria below.
  Interventions: Drug: Aripiprazole Mid (6 - 12 mg/day)
- High (24 - 30 mg/day) (Experimental): Subjects in the 24-30 mg/day group will be administered 2, 6, 12, 18 mg sequentially, each dose once daily for 2 days respectively, followed by a maintenance dose of 24 mg for 34 days. From Day 15 onwards, the dose may be increased to 30 mg in accordance with the criteria below.
  Interventions: Drug: Aripiprazole High (24 - 30 mg/day)

INTERVENTIONS:
Drug: Aripiprazole Low (2 mg/day) — administered 2 mg once daily for 6 weeks
  Other Names: Aripiprazole
  Arms: Low (2 mg/day)
Drug: Aripiprazole Mid (6 - 12 mg/day) — administered 2 mg once daily for 2 days, followed by a maintenance dose of 6 mg for 40 days. From Day 15 onwards, the dose may be increased to 12 mg
  Other Names: Aripiprazole
  Arms: Mid (6 - 12 mg/day)
Drug: Aripiprazole High (24 - 30 mg/day) — administered 2, 6, 12, 18 mg sequentially, each dose once daily for 2 days respectively, followed by a maintenance dose of 24 mg for 34 days. From Day 15 onwards, the dose may be increased to 30 mg
  Other Names: Aripiprazole
  Arms: High (24 - 30 mg/day)

SUMMARY:
The objective of this study is to investigate the efficacy and safety of three different doses of aripiprazole (2 mg/day, 6-12 mg/day, 24-30 mg/day) orally administered over a period of 6 weeks in pediatric patients (aged 13-17 years) with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia (295.30, 295.10, 295.20, 295.90, 295.60), according to DSM-Ⅳ-TR (M.I.N.I.KID will be used as backup)
* Male and female patients aged 13-17 years (between IC and end of dosing)
* Patients with a PANSS score of 70 or more [both at start of dosing (Day 1 and at baseline
* Patients who, in addition to their legal guardian, provide written informed consent, having understood the details of this study
* Inpatient or outpatient status

Exclusion Criteria:

* Patients who have a diagnosis of any other disease except schizophrenia, according to DSM-IV-TR
* Patients who have been compulsorily admitted to hospital
* Patients with mental retardation
* Patients with thyroid disorder
* Patients who have a history of receiving treatment with clozapine, or who have received sufficient doses of two or more kinds of antipsychotic drug for more than four weeks but failed to respond to this treatment
* Patients who have received a prohibited concomitant medication or therapy listed in table 6.4-1 after the start of the prohibited concomitant medication timeframe [to be confirmed at start of dosing (Day 1) and at baseline].
* Patients who have a history of receiving treatment with aripiprazole
* Patients who fall under a contraindication listed in the ABILIFY package insert
* Patients with a serious hepatic, renal, cardiac or hematopoietic disorder
* Patients with a history or a complication of organic brain disorder or convulsive disorder such as epilepsy
* Patients with diabetes. and patients who fall under any of the following:

fasting blood glucose level ≧126 mg/ｄL, non-fasting blood glucose level ≧200 mg/dL, HbA1c≧6.5%

* Patients with a history or a complication of suicide attempt, suicidal thought or self-harm
* Patients with a score of ≧2(mild) on PART1 evaluation of CGI-SS
* Patients with a history or a complication of malignant syndrome, tardive dyskinesia or paralytic ileus
* Patients in a state of physical exhaustion accompanied by such conditions as dehydration or malnutrition
* Patients with a history or a complication of water intoxication
* Patients with Parkinson's disease
* Pregnant women, parturient women, nursing women, women of childbearing potential who wish to become pregnant during this trial. However, women of childbearing potential who are practicing an appropriate method of contraception and have a negative pregnancy test result are eligible for inclusion in this study.
* Patients who have a diagnosis of a substance-related disorder according to DSM-Ⅳ-TR within the past 3 months
* Patients with a positive drug screen (urine) result
* Study enrollment is otherwise judged to be inappropriate by the Investigator or Subinvestigator

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low (2 mg/Day) | Mid (6 - 12 mg/Day) | High (24 - 30 mg/Day)
Started | 35 | 30 | 41
Completed | 27 | 24 | 35
Not Completed | 8 | 6 | 6
Not completed — Adverse Event | 1 | 2 | 5
Not completed — Physician Decision | 3 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low (2 mg/Day) | Mid (6 - 12 mg/Day) | High (24 - 30 mg/Day) | Total
Number analyzed (Participants) | 35 | 30 | 41 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 30 | 41 | 106
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.4) | 15.4 (1.3) | 14.7 (1.3) | 15.0 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 11 | 23 | 55
  Male | 14 | 19 | 18 | 51
Region of Enrollment [Number; unit: participants]
  Japan | 35 | 30 | 41 | 106

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline at Final Assessment in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a 30-item scale where each symptom is rated on a severity scale ranging from 1-7: 1 =Absent, 2 =Minimal, 3 =Mild, 4 =Moderate, 5 =Moderate severe, 6 =Severe, 7= Extreme. PANSS total score is calculated by adding score of 30 items, which ranges from 30-210. Higher scores indicate worse condition.
Time Frame: Baseline (Day 1) and Day 43
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low (2 mg/Day) | Mid (6 - 12 mg/Day) | High (24 - 30 mg/Day)
Number analyzed (Participants) | 35 | 30 | 41
units on a scale | -19.6 (3.2) | -16.5 (3.5) | -21.6 (3.0)

2. Secondary Outcome: Mean Change From Baseline at Final Assessment in Positive and Negative Syndrome Scale (PANSS) Positive Subscale Total Score
Description: The Positive and Negative Syndrome Scale (PANSS) positive subscale score is the sum of the 7 positive item scores (ie, delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution and hostility) and ranges from 7 to 49, with higher values indicating worse condition.
Time Frame: Baseline (Day 1) and Day 43
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low (2 mg/Day) | Mid (6 - 12 mg/Day) | High (24 - 30 mg/Day)
Number analyzed (Participants) | 35 | 30 | 41
units on a scale | -5.2 (0.8) | -4.9 (0.9) | -5.8 (0.8)

3. Secondary Outcome: Mean Change From Baseline at Final Assessment in Clinical Global Impression-Severity of Illness (CGI-S) Score
Description: The Clinical Global Impression-Severity of Illness (CGI-S) Score is a clinician rated scale which assesses how mentally ill the patient is at the time. Scores range from 0 to 7: 0 = Not assessed, 1= Normal, not at all ill, 2 =Borderline mentally ill, 3= Mildly ill, 4= Moderately ill, 5= Markedly ill, 6= Severely ill, 7= Among the most extremely ill patients. Higher scores indicate worse condition.
Time Frame: Baseline (Day 1) and Day43
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low (2 mg/Day) | Mid (6 - 12 mg/Day) | High (24 - 30 mg/Day)
Number analyzed (Participants) | 35 | 30 | 41
units on a scale | -0.9 (0.2) | -0.8 (0.2) | -1.0 (0.2)

4. Secondary Outcome: Mean Change From Baseline at Final Assessment in Clinical Global Impression-Improvement (CGI-I) Score
Description: The Clinical Global Impression-Improvement (CGI-I) Score is a clinician rated scale which assesses the total improvement of the patient's condition compared to that at baseline. Scores range from 0 to 7: 0 = Not assessed, 1= Very much improved, 2 = Much improved, 3= Minimally improved, 4= No change, 5= Minimally worse, 6= Much worse, 7= Very much worse. Higher scores indicate worse condition.
Time Frame: Baseline (Day 1) and day43
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low (2 mg/Day) | Mid (6 - 12 mg/Day) | High (24 - 30 mg/Day)
Number analyzed (Participants) | 35 | 30 | 41
units on a scale | 3.0 (0.2) | 3.2 (0.2) | 2.7 (0.2)

5. Secondary Outcome: Mean Change From Baseline at Final Assessment in Children's Global Assessment Scale (C-GAS) Score
Description: The Children's Global Assessment Scale (C-GAS) is a rating scale which measures psychological, social and school functioning for children aged 6-17. Scores range from 0 to 100, with higher scores indicating better condition.
Time Frame: Baseline (Day 1) and Day 43
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low (2 mg/Day) | Mid (6 - 12 mg/Day) | High (24 - 30 mg/Day)
Number analyzed (Participants) | 35 | 30 | 41
units on a scale | 10.5 (2.0) | 8.5 (2.1) | 8.6 (1.8)

ADVERSE EVENTS:
Time Frame: From the start date of screening examination to date of the final examination (up to Week 6 at e hours after IMP administration)
Arm/Group | Low (2 mg/Day) | Mid (6 - 12 mg/Day) | High (24 - 30 mg/Day)
Serious Adverse Events (participants affected / at risk) | 0/35 | 2/30 | 2/41
Other Adverse Events (participants affected / at risk) | 29/35 | 28/30 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low (2 mg/Day) (N=35) | Mid (6 - 12 mg/Day) (N=30) | High (24 - 30 mg/Day) (N=41)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low (2 mg/Day) (N=35) | Mid (6 - 12 mg/Day) (N=30) | High (24 - 30 mg/Day) (N=41)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (6)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (4) | 9 (11)
Malaise (General disorders) | 3 (3) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (4)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 4 (8)
Somnolence (Nervous system disorders) | 5 (5) | 6 (6) | 5 (5)
Tremor (Nervous system disorders) | 3 (3) | 3 (3) | 6 (6)
Insomnia (Psychiatric disorders) | 5 (5) | 6 (6) | 7 (7)
Schizophrenia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 4 (5) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No